CLINICAL TRIAL: NCT03804918
Title: Mobile Learning Resources as a Tool for Improving Clinician's Ability to Break Bad News: A Pre-post Mixed Methods Pilot Study
Brief Title: Mobile Learning to Improve Clinician's Ability to Break Bad News
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18SM4947
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Education
Keywords: Healthcare education; Breaking bad news; Digital learning

STUDY DESIGN:
Intervention Model Description: A pre-post mixed methods pilot educational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group: All participants (Experimental): Given access to a selected breaking bad news mobile learning resource (VitalTips application).
  Interventions: Other: VitalTips mobile application

INTERVENTIONS:
Other: VitalTips mobile application — VitalTips is a mobile learning application with learning on breaking bad news. Participants were expected to spend at least three hours using the mobile learning resource, ensuring that the time did not impact on their clinical and academic commitments.

SUMMARY:
Design:

A pre-post mixed methods pilot study. All participants granted access to a breaking bad news mobile learning resource (VitalTips).

Baseline and post-intervention questionnaires, pre- and post-intervention simulated patient encounters, and post-intervention semi-structured interviews.

Objective:

To assess if a selected breaking bad news mobile learning resource can improve the ability of clinicians to break bad news.

Population/Eligibility:

15-20 junior doctors and nurses working within two NHS hospitals trusts and one private hospital in England.

Duration:

25th February 2019 to 8th July 2019.

DETAILED DESCRIPTION:
Purpose:

Digital and mobile learning is at the forefront of healthcare education. Though there is evidence for the use of digital learning for practical skills acquisition, there is little evidence of the use of digital learning for breaking bad news training. This pre-post mixed methods pilot study aimed to address this gap in knowledge by assessing how a mobile learning resource may impact the ability of clinicians to break bad news.

Hypothesis:

The addition of a breaking bad news mobile learning resource to clinical practice improves the confidence and ability of junior doctors and nurses to break bad news.

Study objective:

To assess if a breaking bad news mobile learning resource can improve the confidence and ability of clinicians to break bad news.

Methodology:

Potential participants were sent an invitation and participant information sheet (PIS) via e-mail. Potential participants were given up to two weeks to decide if they wanted to participate, with a reminder sent after one week. Each potential participant was referenced by a participant ID number for confidentiality purposes.

Once potential participants read the PIS and given consent, they were asked to complete a baseline questionnaire to understand their demographics, their previous exposure to breaking bad news (through formal or informal training) and their engagement with digital resources.

Following this, participants were asked to complete a baseline simulated patient encounter (SPE) with a simulated patient (SP) (role-played by an actor) to assess their baseline ability to break bad news. Participants were given a task sheet with a brief history of the SP and what news they needed to deliver. The details and history of the SP was documented on a character sheet for the actor's reference. Each participant was given 15 minutes to complete the SPE which was video-recorded. The SPEs were evaluated against the validated Breaking bad news Assessment Schedule (BAS) mark sheet completed by the chief investigator, actor and an independent assessor (by watching the video footage).

Access to the mobile learning resource was granted following the baseline SPE. The mobile learning resource was the freely available VitalTips mobile application, provided by VitalTalks. Participants were expected to spend at least three hours using the mobile learning resource, ensuring that this time did not impact on their clinical and academic commitments.

Four to six weeks later, participants were asked to complete a second videoed SPE, which was marked as described above. The participants were asked to complete a post-intervention questionnaire to gauge the impact on their clinical practice and their engagement with the mobile resources.

The questionnaires utilised a five-point Likert scale ranking of the user's confidence and agreeability with statements. The questionnaires are novel to this study and were developed using the principles of Kirkpatrick's Model of Learning Evaluation, the Theory of Planned Behaviour and the Technology Acceptance Model, whilst also drawing on the most important curricula competencies derived from the content analysis of a sample of medical and nursing curricula followed by an expert consensus.

Soon after the completion of the post-intervention questionnaire, the participants were asked to participate in a 15-30 minutes semi-structured interview with the chief investigator. The participant was asked about their general impressions of the mobile learning resource, their use of the resource in and outside of the clinical environment, their perception of their ability to break bad news before and after the intervention, their perception of their performance in the SPE and any impact on their practice.

Data handling and confidentiality:

Following consent, participants were referenced by their participant ID number (e.g. MLR001). Their e-mail address was recorded next to their participant ID number, gender, role (i.e. doctor or nurse) and training grade, on an Excel spreadsheet for the purpose of contacting participants as the study progressed. Once their commitment to the study had ended, the e-mail addresses were deleted.

Video recordings from the SPEs were transferred from the recording device to a password protected USB stick referenced by the participant ID followed by SPE1 (baseline) or SPE2 (post-intervention), e.g. MLR001_SPE1. Once the independent reviewer had viewed the video and marked the participant, the video file was destroyed.

Audio files from the interviews was transferred from the recording device onto a password protected computer using a USB stick. Once the transfer was completed, the files were deleted from the USB stick. The transferred files were stored on the password protected computer till the returned transcriptions were checked by the chief investigator. Once the files had been checked, the recordings were deleted.

ELIGIBILITY:
Inclusion Criteria:

* Working and training within NHS England and a private healthcare hospital.
* Junior doctor, pre-certificate of completion of training (of any specialty).
* Junior nurse band 5 to 6 (or equivalent) from any specialty.
* Over the age of 18.
* Able to communicate and write in English.
* Willing to engage with mobile learning resources as an additional task to their clinical role, ensuring their learning does not take time out of their clinical commitments.

Exclusion Criteria:

* Medical and nursing students.
* Clinicians who have completed their training programmes i.e. medical or nursing consultants, matrons.
* Retired clinicians.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gehan B Soosaipillai, BM BSc, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - Bupa Cromwell Hospital, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
IPD was only be available on a password protected computer with sole access to the chief investigator. Only anonymised data was sent to the academic supervisor and other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional Group: All Participants: Given access to a selected breaking bad news mobile learning resource (VitalTips application).
  VitalTips mobile application: VitalTips is a mobile learning application with learning on breaking bad news. Participants were expected to spend at least three hours using the mobile learning resource, ensuring that this time does not impact on their clinical and academic commitments.
Period: Overall Study
Arm/Group | Interventional Group: All Participants
Started | 17
Completed | 16
Not Completed | 1
Not completed — Participant did not use the app | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Group: All Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16
Specialty [Count of Participants; unit: Participants]
  Intensive care | 1
  Medicine | 5
  Oncology | 7
  Paediatrics | 1
  Surgery | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-assessed Likert Scale Relating to Confidence in Breaking Bad News at Baseline and Post-intervention.
Description: Baseline and post-intervention questionnaires utilise a five-point Likert scale ranking of the user's confidence and agreeability with statements (Scale: Not very confident at all; Not very confident; Somewhat confident; Very confident; Extremely confident). With each participant acting as their own control, comparisons were made from their own baseline and post-intervention Likert scale ratings.
Time Frame: Baseline questionnaire (week 0) followed by post-intervention questionnaire (weeks 4 to 6)
Population: All participants (n=16) completed both the pre- and post-intervention questionnaires and there was no missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Group: All Participants
Number analyzed (Participants) | 16
Participants
  Pre-intervention: Not very confident at all | 1
  Post-intervention: Not very confident at all | 0
  Pre-intervention: Not very confident | 1
  Post-intervention: Not very confident | 0
  Pre-intervention: Somewhat confident | 12
  Post-intervention: Somewhat confident | 13
  Pre-intervention: Very confident | 2
  Post-intervention: Very confident | 3
  Pre-intervention: Extremely confident | 0
  Post-intervention: Extremely confident | 0

2. Primary Outcome: Change in Simulated Patient Encounter Marking Scores Related to Breaking Bad News at Baseline and Post-intervention.
Description: The simulated patient encounter (SPE) was marked by three assessors using the validated Breaking bad news Assessment Schedule (BAS). The BAS comprises of five sections which group a set of skills relating to BBN. Each skill was marked on a Likert scale in the form of a numerical scale: definitely (positive) 5 _ 4 _ 3 _ 2 _ 1 not at all (negative). The five sections were: A. Setting the scene (minimum score 3; maximum score 15); B. Breaking the news (minimum score 5; maximum score 25); C. Eliciting concerns (minimum score 3; maximum score 15); D. Information giving (minimum score 4; maximum score 20); E. General considerations (minimum score 8; maximum score 40). Overall score (minimum score 23; maximum score 115). Scores from three markers were summed and a mean average was taken pre- and post-intervention for each section and overall. Paired sample t-test were used for analysis of aggregated scores s they enabled the comparison of means between pre- and post-intervention mean scores.
Time Frame: Baseline SPE (week 0) followed by post-intervention SPE (weeks 4 to 6)
Population: All participants (n=16) completed both the pre- and post-intervention SPEs and there was no missing data.
Measure: Mean (Standard Deviation); unit: score on the BAS scale
Arm/Group | Interventional Group: All Participants
Number analyzed (Participants) | 16
score on the BAS scale
  Pre-intervention: Setting the scene | 10.15 (2.54)
  Post-intervention: Setting the scene | 12.25 (1.51)
  Pre-intervention: Breaking the news | 13.31 (5.06)
  Post-intervention: Breaking the news | 20.85 (2.66)
  Pre-intervention: Eliciting concerns | 7.71 (2.54)
  Post-intervention: Eliciting concerns | 10.77 (1.8)
  Pre-intervention: Information giving | 13.23 (2.92)
  Post-intervention: Information giving | 17.46 (1.33)
  Pre-intervention: General considerations | 26.54 (6.08)
  Post-intervention: General considerations | 33.58 (3.72)
  Pre-intervention: Overall | 71.15 (17.19)
  Post-intervention: Overall | 94.92 (9.58)

ADVERSE EVENTS:
Time Frame: AE data was not collected due to it being an observational study and no AE's were anticipated.
Description: No AE's were expected and AE's were not monitored for this reason.
Arm/Group | Interventional Group: All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Sample numbers were small, which affects the interpretation of the quantitative measures (BAS mark sheet). Participants learned both from the app and the SPEs. Any change in the skill set must also take into consideration the learning from the SPEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT03804918/Prot_SAP_ICF_000.pdf